CLINICAL TRIAL: NCT01872156
Title: Effectiveness of an Intervention in Primary Care to Promote Smoking Cessation in Pregnant Women: Cluster Randomized Controlled Trial.
Brief Title: Effectiveness of an Intervention in Primary Care to Promote Smoking Cessation in Pregnant Women
Acronym: GESTABAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOMAMFYC11/2012
Record Dates: First submitted 2013-04-24; First posted 2013-06-07 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Cessation, Smoking
Keywords: Smoking; Primary care
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention GESTABAC (Experimental): Intervention based on the "Clinician's Guide to helping Pregnant Women Quit Smoking" on the rates of abstinence of the patients in whom it has been controlled in this period of time, at the end of the pregnancy and after the childbirth.
  Interventions: Other: Intervention GESTABAC
- Control Group (Other): The group control will act according to usual management.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention GESTABAC — Intervention based on the "Clinician's Guide to helping Pregnant Women Quit Smoking" on the rates of abstinence of the patients in whom it has been controlled in this period of time, at the end of the pregnancy and after the childbirth.
  Arms: Intervention GESTABAC
Other: Control Group — The group control will act according to usual management.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the behavior treatment accompanied by self-help materials in Primary health care, across the intervention of the midwifes in the pregnancy follow-up visits.

DETAILED DESCRIPTION:
Aim: To evaluate the efficiency of an intervention in smoking based on a clinical practice guideline on the part of the primary care professionals on tobacco abstinence at the conclusion of the pregnancy self referred and validated with cooximetry.

Secondary objectives:

1. To evaluate the effectiveness of an intervention in smoking based on a clinical practice guideline on the part of the primary care professionals on the tobacco abstinence 6 months after the childbirth.
2. The effectiveness of the intervention values on the weight of the newborn child, the number of childbirths pre-term and the perinatal mortality.
3. To study the effectiveness of the intervention in smoking on the maintenance of the breast-feeding to 3 and 6 months.

Method:

Design: cluster randomized controlled trial. Setting: study in Health Centers Primary Care of Area of Madrid Health Service.

Sample size adjusted for design effect: number of smoking women in every branch would be of 350.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* pregnant at 20 weeks or less of gestation
* attending her first prenatal visit with any of the participating prenatal care teams (this first prenatal visit takes place usually around 6-12 weeks of pregnancy)
* defining herself as a current cigarette smoker or recent ex-smoker (see below for a definition of these terms)
* being able to meet the requisites of the trial:
* being available for the next 15 months
* defining herself as fluent in reading and speaking Spanish to understand the study procedures and to comply with them

  * meeting no exclusion criterion; and
  * willing and able to give informed consent for participation in the study

Exclusion Criteria:

* communication barrier;
* active addictions to other psychoactive substances
* involved in any other formal smoking cessation program or in another trial during the study period; or
* does not consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Rate of abstinence of tobacco | 6 months
  Rate of abstinence of tobacco to 20-28 weeks of childbearing , to 36-38 weeks and to 6 postpartum (post-childbearing) months. The abstinence will be validated for cooximetry.

CONTACTS AND LOCATIONS:
Overall Officials: Encarnación Serrano-Serrano, MD, Principal Investigator — Gerencia de Atención Primaria, Madrid
Locations (1):
- Gerencia de Atención Primaria, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: An online platform to facilitate communication and dissemination of information between the research group — http://gestabac.wordpress.com